CLINICAL TRIAL: NCT02470910
Title: Incorporating MR Imaging Into Prostate Radiotherapy Treatment Planning: A Pilot Study to Quantitate the Potential to Limit Radiation Dose to Normal Tissues.
Brief Title: Incorporating MR Imaging Into Prostate Radiotherapy Treatment Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Anthony V. D'Amico, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-585
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate Stage I; Adenocarcinoma of the Prostate Stage II; Adenocarcinoma of the Prostate Stage III
Keywords: Prostate Cancer; Stage I-III prostate adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic resonance imaging (Experimental): MRI examination after intraprostatic fiducial markers have been placed and prior to beginning radiotherapy
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging
  Other Names: MRI

SUMMARY:
This research study is evaluating whether a standard prostate MRI examination can improve radiation therapy planning for prostate cancer.

DETAILED DESCRIPTION:
In this research study, the investigators want to determine if prostate radiotherapy treatment planning can be improved by using an MRI scan to help doctors more accurately target the prostate with radiation and decrease radiation dose to the rectum, which is just behind the prostate.

To do this, the investigators will create a treatment plan based on the MRI scan and compare it to the standard treatment, which currently uses a CT scan rather than an MRI. The results of this study will help inform doctors whether it is beneficial to routinely use an MRI scan for prostate radiotherapy treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed prostate cancer.
* PSA level and prostate biopsy must be reviewed at Brigham and Women's Hospital or the Dana Farber Cancer Institute and should support a diagnosis of stage I-III prostate adenocarcinoma.
* Candidates with PSA greater than 20, digital rectal exam consistent with disease outside the prostate (clinical T3/T4 disease), or Gleason score 8 or greater, should have a bone scan and diagnostic pelvic CT or MRI to exclude metastatic disease.
* Prostate biopsy, serum PSA measurement, and any indicated diagnostic imaging studies must be performed within 60 days of the date of registration.
* Participants should not have had prior curative local treatment for prostate cancer, including no radiotherapy or prostatectomy. A maximum 90 days of systemic androgen deprivation therapy prior to registration is allowed.
* Participation is limited to adult patients, age 18 years or older.
* ECOG performance status ≥2 (Karnofsky ≥60%)
* Life expectancy of greater than 10 years.
* Able to tolerate an MRI examination.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with known or suspected metastatic (stage IV) prostate cancer.
* Participants with an implanted device, prosthesis, or any other foreign body with ferromagnetic properties that would make them ineligible to undergo MRI examination.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D'Amico, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kuban DA, Levy LB, Cheung MR, Lee AK, Choi S, Frank S, Pollack A. Long-term failure patterns and survival in a randomized dose-escalation trial for prostate cancer. Who dies of disease? Int J Radiat Oncol Biol Phys. 2011 Apr 1;79(5):1310-7. doi: 10.1016/j.ijrobp.2010.01.006. Epub 2010 May 20. PMID 20493642
- [Background] Zietman AL, Bae K, Slater JD, Shipley WU, Efstathiou JA, Coen JJ, Bush DA, Lunt M, Spiegel DY, Skowronski R, Jabola BR, Rossi CJ. Randomized trial comparing conventional-dose with high-dose conformal radiation therapy in early-stage adenocarcinoma of the prostate: long-term results from proton radiation oncology group/american college of radiology 95-09. J Clin Oncol. 2010 Mar 1;28(7):1106-11. doi: 10.1200/JCO.2009.25.8475. Epub 2010 Feb 1. PMID 20124169
- [Background] Sanda MG, Dunn RL, Michalski J, Sandler HM, Northouse L, Hembroff L, Lin X, Greenfield TK, Litwin MS, Saigal CS, Mahadevan A, Klein E, Kibel A, Pisters LL, Kuban D, Kaplan I, Wood D, Ciezki J, Shah N, Wei JT. Quality of life and satisfaction with outcome among prostate-cancer survivors. N Engl J Med. 2008 Mar 20;358(12):1250-61. doi: 10.1056/NEJMoa074311. PMID 18354103
- [Background] Debois M, Oyen R, Maes F, Verswijvel G, Gatti G, Bosmans H, Feron M, Bellon E, Kutcher G, Van Poppel H, Vanuytsel L. The contribution of magnetic resonance imaging to the three-dimensional treatment planning of localized prostate cancer. Int J Radiat Oncol Biol Phys. 1999 Nov 1;45(4):857-65. doi: 10.1016/s0360-3016(99)00288-6. PMID 10571190
- [Background] Rasch C, Barillot I, Remeijer P, Touw A, van Herk M, Lebesque JV. Definition of the prostate in CT and MRI: a multi-observer study. Int J Radiat Oncol Biol Phys. 1999 Jan 1;43(1):57-66. doi: 10.1016/s0360-3016(98)00351-4. PMID 9989514
- [Background] Roach M 3rd, Faillace-Akazawa P, Malfatti C, Holland J, Hricak H. Prostate volumes defined by magnetic resonance imaging and computerized tomographic scans for three-dimensional conformal radiotherapy. Int J Radiat Oncol Biol Phys. 1996 Jul 15;35(5):1011-8. doi: 10.1016/0360-3016(96)00232-5. PMID 8751410
- [Background] Parker CC, Damyanovich A, Haycocks T, Haider M, Bayley A, Catton CN. Magnetic resonance imaging in the radiation treatment planning of localized prostate cancer using intra-prostatic fiducial markers for computed tomography co-registration. Radiother Oncol. 2003 Feb;66(2):217-24. doi: 10.1016/s0167-8140(02)00407-3. PMID 12648794
- [Derived] Schmidt DR, Bhagwat M, Glazer DI, Chen MH, Moteabbed M, McMahon E, Loffredo MJ, Tempany CM, D'Amico AV. MRI-Based Radiotherapy Planning to Reduce Rectal Dose in Excess of Tolerance. Prostate Cancer. 2022 Feb 3;2022:7930744. doi: 10.1155/2022/7930744. eCollection 2022. PMID 35154830

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnetic Resonance Imaging: Magnetic Resonance Imaging (MRI) examination after intraprostatic fiducial markers have been placed and prior to beginning radiotherapy.
Period: Overall Study
Arm/Group | Magnetic Resonance Imaging
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Magnetic Resonance Imaging: MRI examination after intraprostatic fiducial markers have been placed and prior to beginning radiotherapy
  Magnetic Resonance Imaging
Arm/Group | Magnetic Resonance Imaging
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 70 [56 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Rectal Volume Receiving 70 Gy or More With CT Versus MRI-planned Prostate Radiotherapy.
Description: The volume of rectum receiving or exceeding 70 Gy will be calculated from the dose-volume histogram. Results will be compared for CT and MRI-based plans.
Time Frame: within 1 year of MRI examination
Measure: Median (Inter-Quartile Range); unit: cubic centimeters
Groups:
- MRI-based Planning: A radiation therapy plan was designed using MRI-defined prostate volume. Median volume of rectum receiving 70Gy or more was calculated from the dose-volume histogram.
- CT-based Planning: A radiation therapy plan was designed using CT-defined prostate volume. Median volume of rectum receiving 70Gy or more was calculated from the dose-volume histogram.
Arm/Group | MRI-based Planning | CT-based Planning
Number analyzed (Participants) | 15 | 15
cubic centimeters | 4.9 [4.1 to 8.7] | 9.3 [7.0 to 10.2]

2. Secondary Outcome: Comparison of Bladder Volume Receiving 70 Gy or More With CT Versus MRI-planned Prostate Radiotherapy.
Description: The volume of bladder receiving or exceeding 70 Gy will be calculated from the dose-volume histogram. Results will be compared for CT and MRI-based plans.
Time Frame: within 1 year of MRI examination
Measure: Median (Inter-Quartile Range); unit: cubic centimeters
Groups:
- MRI-based Planning: A radiation therapy plan was designed using MRI-defined prostate volume. Median volume of bladder receiving 70 Gy or more was calculated from the dose-volume histogram.
- CT-based Planning: A radiation therapy plan was designed using CT-defined prostate volume. Median volume of bladder receiving 70 Gy or more was calculated from the dose-volume histogram.
Arm/Group | MRI-based Planning | CT-based Planning
Number analyzed (Participants) | 15 | 15
cubic centimeters | 9.6 [8.2 to 12.9] | 12.7 [10.8 to 15.0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Magnetic Resonance Imaging
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT02470910/Prot_SAP_000.pdf